CLINICAL TRIAL: NCT04140435
Title: How Does the EUS-guided Through-the-needle Microforceps Biopsy Improve Diagnosis of Pancreatic Cystic Lesions: A Multicenter Prospective Study
Brief Title: EUS-guided Through-the-needle Microforceps Biopsy Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Gastroenterology and Advance Endoscopy (Other)
Responsible Party: Sponsor
Other Study IDs: IGEA07-2019
Record Dates: First submitted 2019-10-22; First posted 2019-10-25 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Pancreatic Cyst
Keywords: EUS-guided through the needle biopsy (EUS-guided TTNB); Pancreatic cyst lesions (PCLs)
MeSH Terms: conditions — Pancreatic Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples of cyst wall
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TTNB group: Patients with PCLs suitable for biopsy.
  Interventions: Device: EUS-guided through-the-needle microbiopsy forceps (Moray)

INTERVENTIONS:
Device: EUS-guided through-the-needle microbiopsy forceps (Moray) — EUS-TTNB procedure technique. An endosonographer of each institution will perform the EUS procedures. Cysts morphology will be recorded and then punctured by using a 19-gauge EUS-FNA needle. Then the through-the-needle microbiopsy forceps (Moray) will be inserted through the needle into the cystic lumen. Microbiopsies will be obtained from the cyst wall randomly and from mural nodules or septae when observed. The open jaws of the forceps will be pushed onto the cyst wall, closed and pulled back to cause visible tenting. Two "bites" per pass will be obtained. Then the forceps will be removed and the specimen placed in formalin vials. The procedure will be repeated 2 times, or until 2 visible specimens are obtained. After completion of biopsies, the cyst fluid will be completely aspirated and sent for CEA, amylase, glucose and cytology analyses. If a mural nodule is visualized on EUS, it will be accessed separately by using the 19-gauge needle for EUS-FNA cytology.

SUMMARY:
INTRODUCTION: The diagnosis of pancreatic cystic lesions (PCLs) is increasing due to improvements of cross-sectional imaging. It is mandatory, for appropriate management, to make an accurate diagnosis and risk stratification, since some of these lesions may harbor malignancy or have potential for malignant transformation and hence surgical resection is required. Diagnostic evaluation of PCLs can be challenging, requiring a combination of different methods. Usually PCLs are been initially detected by cross-sectional imaging. However, imaging alone has not been shown to reliably identify the underlying pathology in PCLs with a high degree of accuracy. Hence, Endoscopic ultrasound with fine-needle aspiration (EUS-FNA) is routinely performed. EUS-FNA plays an important role in cyst characterization since allows morphological examination (EUS-B mode), aspiration for cytology and cyst fluid analysis for carcinoembryonic antigen (CEA), amylase and glucose levels; and allows to tissue sample in case of mural nodules o wall thickness. Even though EUS-FNA has been shown to be the test of choice for select lesions with high-risk features, has its limitations related to low sensitivity and specificity. The morphological characterization by EUS of PCL, as well as with the cross-sectional images, depends most of the time, on the subjective interpretation of the operator, which can be very difficult sometimes and depend on experience. A cyst fluid CEA cutoff of 192 ng/mL has been commonly accepted for differentiating mucinous from non-mucinous cysts. However, has the limitation of requiring at least 0.5 mL of cyst fluid for CEA analysis, has a relatively low sensitivity (75%) and specificity (84%), cannot differentiate cyst histotypes, and controversial results have been reported. Finally targeted cyst wall with the tip of the FNA needle can increase the diagnostic accuracy, yet the cytological yield with EUS-FNA remains low due to the relatively small tissue sample. Hence, diagnostic accuracy of currently available tools for evaluation of PCLs including cross-sectional imaging, EUS morphologic features, EUS-FNA for cyst fluid analysis and cytology is not perfect, leading to possible misdiagnosis.

DETAILED DESCRIPTION:
Recently, a EUS-guided through-the-needle microforceps device (Moray Micro Forceps, US Endoscopy, Mentor, Ohio, United States), witch can be passed through the lumen of a 19-gauge FNA needle, has been introduced as a novel approach for PCLs tissue acquisition. It has been shown that this device can drastically changed the diagnosis, providing diagnoses otherwise not suggested by cytology or cyst fluid CEA levels. The possibility of obtaining histological specimens from the cyst wall with this microforceps may change the management os PCLs, by obtening enough material for supplementary immunohistochemical analysis, allowing for even more accurate histological diagnosis, and in the case of IPMNs, possibly histological subtyping. The aims of this study is to assess: 1) the increment in diagnostic yield, by using this device, when compared to standard evaluation with cross-sectional imaging, EUS-FNA with cyst fluid analysis, 2) to evaluate the technical success, clinical success and safety, 3) Finally inter-observer accuracy in the assessment of PCLs using the different methods will be mesure, by the participation of all the endosonographers of Argentina, in the context of the annual EUS meeting.

• MATERIALS AND METHODS Study design and Setting: It is multicenter, prospective, interventional, non-controlled or randomized and double blind study, performed at the Institute of Gastroenterology and Advanced Endoscopy - IGEA (Bahía Blanca, Argentina), in conjunction with five high volume centers of all over Argentina (La Plata, Buenos Aires x 2, Neuquen and Mendoza), with patients included from July 2019 to July 2020. The study protocol and consent form has been approved by the institutional review board, will be registered at ClinicalTrials.gov and will be conducted according to the declaration of Helsinki. Written informed consent will be obtained from all subjects. No financial support will be received from the manufacturer of the microforceps, and none of the authors have any conflicts of interest. Data collection: Patient demographics, clinical history, cross-sectional imaging and EUS cyst findings like number of cysts, location, size and features (unilocular/septated, mural nodules, thickened wall, communication with pancreatic duct, dilated pancreatic duct and solid component) will be review. Fluid characteristics (viscosity, color, volume), amylase, glucose, CEA level and citology will be analyzed. The CEA level will be classified as <5, 6-192, >192 ng/mL and glucose level as > 50 and ≤ 50 mg/dl. ( ) EUS-FNA type of needle used, biopsy route (stomach/duodenum) and number of passes will be recorded as well as TTNB number of biopsies. Adverse events, technical and clinical success of EUS-FNA and TTNB will be recorded. Results of both procedures will be expressed in terms of cyst histotype, grade of dysplasia and mucinous vs. nonmucinous. Finally surgery result and follow up (12 month) will be used as gold standards. Follow-up data will be obtained from clinical encounters and/or telephone calls. Adverse events will be recorded per published American Society for Gastrointestinal Endoscopy criteria. Intervention: EUS-TTNB procedure technique. All procedures will be performed in a hospital-based interventional endoscopy suite, under intravenous sedation in a standardized manner and under antibiotics prophylactic. In cases of intracystic bleeding or impossibility of emptying the cyst, antibiotic therapy will be prolonged for 5 days. An endosonographer of each institution will perform the EUS procedures, but all the endosonographers of Argentina will analyze the results. EUS procedures will be performed with a linear echo-endoscope (EG-3870 UTK - Pentax, Tokyo, Japan; Hitachi Medical Systems, Tokyo, Japan). Cysts morphology will be recorded as was previously described and then punctured under Doppler guidance by using a 19-gauge EUS-FNA needle (Expect needle; Boston Scientific, Marlborough, Mass or EchoTip Ultra needle; Cook Medical, Bloomington, Ind). The stylet will be removed and the through-the-needle microbiopsy forceps (Moray; US Endoscopy, Mentor, Ohio, USA), with a sheath diameter of 0.8 mm and a jaw opening width of 4.3 mm, will be inserted through the needle into the cystic lumen. Microbiopsies will be obtained from the cyst wall randomly and from mural nodules or septae when observed. The open jaws of the forceps will be pushed gently onto the cyst wall, closed and pulled back to cause visible tenting. Two "bites" per pass of the microforceps will be obtained. Then the forceps will be removed, leaving the needle tip inside the cyst, the specimen will be placed in formalin vials and the forceps will be generously washed with normal saline solution before repeat biopsy. In the absence of intracystic bleeding, the procedure will be repeated 2 times, based on previous information with this device, or until 2 visible specimens are obtained. After completion of biopsies, the cyst fluid will be completely aspirated and sent for biochemistry (CEA, amylase, glucose) and cytology analyses, as was previously mentioned. If the cyst fluid is scarce, analysis of CEA concentration will be preferred over cytology. If a mural nodule is visualized on EUS, it will be accessed separately by using the 19-gauge needle for EUS-FNA cytology. No on-site cytopathological examination will be performed and all specimens will be evaluated by experienced gastrointestinal cytopathologists. Microbiopsies will be fixed immediately in 10% formalin solution and send to be stained with standard hematoxylin and eosin (H and E) and supplementary immunohistochemical (IHC) staining when indicated. After the procedure, patients will be observed for 2 hours in the recovery room before being discharged.

Definitions: Technical success will be defined as successful puncture of the pancreatic cyst with the 19-gauge needle under EUS guidance, advance the microforceps into the cyst, and successful tissue acquisition, that will be confirmed by gross visualization of the specimen from the jaws of the forceps. Clinical success will be defined as the ability to obtain a histopathological diagnosis of the PCL, by cytological or histological evaluation, using the microforceps biopsies. TTNB specimen diagnostic accuracy will be calculated at 3 different diagnostic levels: 1) Provide a specific diagnosis of the cyst histotype based on the characteristics of the epithelium and/or the cells composing the cyst wall. 2) Define the grade of dysplasia. 3) Differentiate mucinous versus nonmucinous cysts based on: The presence of a mucinous epithelium with cytoplasmic mucin and the presence of colloid-like extracellular mucin. The TTNB sampling diagnostic reliability (sensitivity and specificity) will be assessed by the evaluation of the correlation between the TTNB sampling results and surgical specimens (Gold Standard) in patients who underwent surgery or 12 months follow up in case of non-surgical PCL. Cysts with characteristics consistent with mucinous pancreatic cystic (mucinous epithelium with cytoplasmic mucin and/or colloid-like extracellular mucin) on FNA cytology, microforceps histology and/or surgical histology (when available) will be determined as mucinous pancreatic cystic. Otherwise, a final diagnosis will be determined, based on available cross-section imaging, EUS characterization, cyst fluid markers (CEA≥ 192 ng/mL and glucose ≤ 50) and stable appearance on 12 months follow-up. Cyst fluid CEA will be used to initially categorize the lesion as likely non-mucinous (CEA< 192 ng/mL), likely mucinous (CEA≥ 192 ng/mL) or inconclusive (between 6 and 191 ng/mL). Adverse events (AEs) will be defined and classified according to American Society for Gastrointestinal Endoscopy guidelines. Interobserver Agreement: It was mentioned before that diagnostic evaluation of PCLs can be challenging, requiring a combination of different methods, that many of them may have a low sensitivity and specificity, being dependent most of the time, on the subjective interpretation of the operator, which can be very difficult sometimes and experience dependent. The increment in diagnostic yield of a new method is appreciated as the result of the comparison of the new and previous methods accuracy. It is rational to understand that, if the method accuracy is experience dependent, this difference between methods accuracy will be less in more experience work groups. So when the increment in diagnostic yield of a new procedure is been analyzed it is important to ensure that the results can be apply to most of the practitioners (external validity/inter-observer agreement) and not only one group of work since it will only reflect the experience of that group (internal validity/ intra-observer agreement). For that outcome is that inter-observer agreement will be evaluated in the context of the Argentinian annual EUS meeting, where different cases will be presented to all the endosonographers of Argentina. Cases will be presented in 3 stages where a diagnostic assessment will have to be made in each stage. Initially (1st stage) patient's demographic data (sex, age), clinical history and images (CT, MRI, ultrasound) will be shown. Then (2nd stage) EUS images and videos will be presented and finally (3rd stage) the cyst fluid analysis results biochemistry (CEA, glucose, amylase) and cytology will be reviewed. Only 10 cases will be analyzed, during the meeting, due to time limitation, and agreement will be continue beeing evaluated using an online platform where cases will be presented using the same methodology. An external assistant to the protocol will analyze all the result and the different institutes will provide the cases, in a double blind manner, where neither the participating physician nor the operators will know the final results (TTNB or surgery).

Statistical analysis: Summary data will be expressed as mean +/- standard deviation (SD), or median and range for continuous variables and as number with percentage for categorical variables. Fisher o Chi-square test for categorical variables and the t test for continuous variables will be performed when indicated. The sensitivity, specificity, predictive values and accuracy of TTNB will be calculated with the 95% Confidence Interval (95% CI). To examine inter-observer agreement, kappa values will be calculated. Kappa coefficients below 0.4 indicate "poor agreement," values between 0.4 and 0.8 represent "moderate to good agreement," and values greater than 0.8 indicate "excellent agreement." A P value < 0.05 will be considered to be statistically significant. All the statistical analysis will be performed using SPSS software suite v.22.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old patients.
* Patints that agree to participate in the study.
* PCLs ≥ 10mm, large enough to accommodate the microforceps.
* Patients with PCLs and high-risk features (cyst > 3 cm, thickened wall, dilated pancreatic duct, mural nodules and solid component).
* New diagnosis of a PCL or interval changes in morphology on surveillance (cyst growth or high-risk features).
* Patients with PCLs and symptoms (e. g. pancreatitis, abdominal pain, obstructive jaundice).
* Patients with PCLs but without high-risk features and anxiety about the diagnosis.

Exclusion Criteria:

* Inability to provide informed consent for the procedure.
* Pregnancy.
* Platelet count less than 50,000/ml or International Normalized Rate (INR) >2.
* Esophageal stricture or any pathology that does noy allows performing EUS.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic cysts suitable for EUS TTNB with microforceps.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
The increment in diagnostic yield | 1 year
  The diagnostic performance (accuracy) of the device will be compared to standard evaluation accuracy (cross-sectional imaging and EUS-FNA with cyst fluid analysis) and finally corroborated with surgery biopsy and 12 month follow up (gold standard).

SECONDARY OUTCOMES:
Percentage of technical success | 1 year
  It will be measured the cases in witch a successful puncture of the pancreatic cyst with the 19-gauge needle under EUS guidance, advance the microforceps into the cyst, and successful tissue acquisition was performed. It will be confirmed by gross visualization of the specimen from the jaws of the forceps.
Percentage of clinical success | 1 year
  It will be measured the cases in witch a histopathological diagnosis of the PCL, by cytological or histological evaluation, using the microforceps biopsies was obtained.
Percentage of adverse events | 1 year
  All adverse events will recorded according to American Society for Gastrointestinal Endoscopy guidelines.
The inter-observer agreement | 1 year
  It will be evaluated if the increment in diagnostic yield can be generalized. All cases will be presented to all the endosonographers of Argentina, in the context of the annual EUS meeting and then by an online platform, where they will have to asses a diagnosis in three stages: 1st stage: patient's demographic data, clinical history and images (CT, MRI, ultrasound). 2nd stage: EUS features (EUS-B mode). 3rd stage: cyst fluid analysis CEA, glucose, amylase and cytology.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Valero, MD, Principal Investigator — Institute of Gastroenterology and Advanced Endoscopy (IGEA)
Locations (1):
- Institute of Gastroenterology and Advanced Endoscopy (IGEA), Bahía Blanca, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stark A, Donahue TR, Reber HA, Hines OJ. Pancreatic Cyst Disease: A Review. JAMA. 2016 May 3;315(17):1882-93. doi: 10.1001/jama.2016.4690. PMID 27139061
- [Result] Lee KS, Sekhar A, Rofsky NM, Pedrosa I. Prevalence of incidental pancreatic cysts in the adult population on MR imaging. Am J Gastroenterol. 2010 Sep;105(9):2079-84. doi: 10.1038/ajg.2010.122. Epub 2010 Mar 30. PMID 20354507
- [Result] Correa-Gallego C, Ferrone CR, Thayer SP, Wargo JA, Warshaw AL, Fernandez-Del Castillo C. Incidental pancreatic cysts: do we really know what we are watching? Pancreatology. 2010;10(2-3):144-50. doi: 10.1159/000243733. Epub 2010 May 17. PMID 20484954
- [Result] Cho CS, Russ AJ, Loeffler AG, Rettammel RJ, Oudheusden G, Winslow ER, Weber SM. Preoperative classification of pancreatic cystic neoplasms: the clinical significance of diagnostic inaccuracy. Ann Surg Oncol. 2013 Sep;20(9):3112-9. doi: 10.1245/s10434-013-2986-6. Epub 2013 Apr 18. PMID 23595223
- [Result] Rogart JN, Loren DE, Singu BS, Kowalski TE. Cyst wall puncture and aspiration during EUS-guided fine needle aspiration may increase the diagnostic yield of mucinous cysts of the pancreas. J Clin Gastroenterol. 2011 Feb;45(2):164-9. doi: 10.1097/MCG.0b013e3181eed6d2. PMID 20818233
- [Result] Hong SK, Loren DE, Rogart JN, Siddiqui AA, Sendecki JA, Bibbo M, Coben RM, Meckes DP, Kowalski TE. Targeted cyst wall puncture and aspiration during EUS-FNA increases the diagnostic yield of premalignant and malignant pancreatic cysts. Gastrointest Endosc. 2012 Apr;75(4):775-82. doi: 10.1016/j.gie.2011.12.015. Epub 2012 Feb 7. PMID 22317883
- [Result] Alkaade S, Chahla E, Levy M. Role of endoscopic ultrasound-guided fine-needle aspiration cytology, viscosity, and carcinoembryonic antigen in pancreatic cyst fluid. Endosc Ultrasound. 2015 Oct-Dec;4(4):299-303. doi: 10.4103/2303-9027.170417. PMID 26643697
- [Result] Brugge WR, Lewandrowski K, Lee-Lewandrowski E, Centeno BA, Szydlo T, Regan S, del Castillo CF, Warshaw AL. Diagnosis of pancreatic cystic neoplasms: a report of the cooperative pancreatic cyst study. Gastroenterology. 2004 May;126(5):1330-6. doi: 10.1053/j.gastro.2004.02.013. PMID 15131794
- [Result] de Jong K, Poley JW, van Hooft JE, Visser M, Bruno MJ, Fockens P. Endoscopic ultrasound-guided fine-needle aspiration of pancreatic cystic lesions provides inadequate material for cytology and laboratory analysis: initial results from a prospective study. Endoscopy. 2011 Jul;43(7):585-90. doi: 10.1055/s-0030-1256440. Epub 2011 May 24. PMID 21611945
- [Result] Gaddam S, Ge PS, Keach JW, Mullady D, Fukami N, Edmundowicz SA, Azar RR, Shah RJ, Murad FM, Kushnir VM, Watson RR, Ghassemi KF, Sedarat A, Komanduri S, Jaiyeola DM, Brauer BC, Yen RD, Amateau SK, Hosford L, Hollander T, Donahue TR, Schulick RD, Edil BH, McCarter M, Gajdos C, Attwell A, Muthusamy VR, Early DS, Wani S. Suboptimal accuracy of carcinoembryonic antigen in differentiation of mucinous and nonmucinous pancreatic cysts: results of a large multicenter study. Gastrointest Endosc. 2015 Dec;82(6):1060-9. doi: 10.1016/j.gie.2015.04.040. Epub 2015 Jun 12. PMID 26077458
- [Result] Mittal C, Obuch JC, Hammad H, Edmundowicz SA, Wani S, Shah RJ, Brauer BC, Attwell AR, Kaplan JB, Wagh MS. Technical feasibility, diagnostic yield, and safety of microforceps biopsies during EUS evaluation of pancreatic cystic lesions (with video). Gastrointest Endosc. 2018 May;87(5):1263-1269. doi: 10.1016/j.gie.2017.12.025. Epub 2018 Jan 6. PMID 29309781
- [Result] Tanaka M, Fernandez-del Castillo C, Adsay V, Chari S, Falconi M, Jang JY, Kimura W, Levy P, Pitman MB, Schmidt CM, Shimizu M, Wolfgang CL, Yamaguchi K, Yamao K; International Association of Pancreatology. International consensus guidelines 2012 for the management of IPMN and MCN of the pancreas. Pancreatology. 2012 May-Jun;12(3):183-97. doi: 10.1016/j.pan.2012.04.004. Epub 2012 Apr 16. PMID 22687371
- [Result] Scheiman JM, Hwang JH, Moayyedi P. American gastroenterological association technical review on the diagnosis and management of asymptomatic neoplastic pancreatic cysts. Gastroenterology. 2015 Apr;148(4):824-48.e22. doi: 10.1053/j.gastro.2015.01.014. No abstract available. PMID 25805376
- [Result] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Result] Crino SF, Bernardoni L, Brozzi L, Barresi L, Malleo G, Salvia R, Frulloni L, Sina S, Parisi A, Remo A, Larghi A, Gabbrielli A, Manfrin E. Association between macroscopically visible tissue samples and diagnostic accuracy of EUS-guided through-the-needle microforceps biopsy sampling of pancreatic cystic lesions. Gastrointest Endosc. 2019 Dec;90(6):933-943. doi: 10.1016/j.gie.2019.05.009. Epub 2019 May 14. PMID 31100310
- [Result] Yang D, Samarasena JB, Jamil LH, Chang KJ, Lee D, Ona MA, Lo SK, Gaddam S, Liu Q, Draganov PV. Endoscopic ultrasound-guided through-the-needle microforceps biopsy in the evaluation of pancreatic cystic lesions: a multicenter study. Endosc Int Open. 2018 Dec;6(12):E1423-E1430. doi: 10.1055/a-0770-2700. Epub 2018 Dec 5. PMID 30574535